CLINICAL TRIAL: NCT07285122
Title: A Phase I, Randomised, Double Blind, Placebo-controlled, Dose-escalating Study of the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of RB042 Administered Via Inhalation to Healthy Adult Volunteers and Healthy Adult Smokers
Brief Title: Inhaled RB042 in Healthy Adult Volunteers and Healthy Adult Smokers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: RAGE Bio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RB042_1001
Record Dates: First submitted 2025-12-03; First posted 2025-12-16 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Healthy; Healthy Smoker

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Cohort A1 (Experimental): Participants will receive RB042 (Dose Level A1) or matching placebo on Day 1.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution
- Cohort A2 (Experimental): Participants will receive RB042 (Dose Level A2) or matching placebo on Day 1.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution
- Cohort A3 (Experimental): Participants will receive RB042 (Dose Level A3) or matching placebo on Day 1.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution
- Cohort A4 (Experimental): Participants will receive RB042 (Dose Level A4) or matching placebo on Day 1.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution
- Cohort B1 (Experimental): Participants will receive RB042 (Dose Level B1) or matching placebo on Days 1, 8, 15, and 22.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution
- Cohort B2 (Experimental): Participants will receive RB042 (Dose Level B2) or matching placebo on Days 1, 8, 15, and 22.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution
- Cohort B3 (Experimental): Participants will receive RB042 (Dose Level B3) or matching placebo on Days 1, 8, 15, and 22.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution
- Cohort C1 (Experimental): Participants will receive RB042 (Dose Level C1) or matching placebo on Days 1, 8, 15, and 22.
  Interventions: Drug: RB042; Drug: Placebo inhalation solution

INTERVENTIONS:
Drug: RB042 — A single or multiple doses of RB042 will be administered via a nebuliser.
Drug: Placebo inhalation solution — A single or multiple doses of placebo will be administered via a nebuliser.

SUMMARY:
This is a 3-part, randomised, double-blind, placebo-controlled, first in human study evaluating the safety, tolerability, pharmacokinetics, and pharmacodynamics of inhaled RB042.

DETAILED DESCRIPTION:
The purpose of this study is to measure the safety, tolerability, PK, and PD of inhaled RB042 compared with inhaled placebo in healthy adult volunteers and healthy adult smokers.

Study details include:

* Overall study duration of up to 14 months.
* Participants in Part A (healthy adult volunteers) will be required to visit the study site for assessments on 11 occasions, including a 4-day in-house stay, over 4 months.
* Participants in Parts B (healthy adult volunteers) and C (healthy adult smokers) will be required to visit the study site for assessments on 13 occasions, including a 17-day (Day -1 to 16) and 3-day (Day 21 to 24) in-house stay, over 5 months.
* Participants will be administered a single dose (Part A) or multiple doses (Parts B and C) of study intervention.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be overtly healthy as determined by medical evaluation
* Part C only: have a ≥10 pack years smoking history, have smoked tobacco products (cigarettes, cigars, or equivalent) regularly for the past 12 months, and currently smoke daily.
* Have forced expiratory volume (FEV1) ≥80% predicted and FEV1 to FVC ratio (FEV1/FVC) ≥0.7 at Screening and on Day -1
* Body weight at least 50 kg and have a body mass index (BMI) within the range 18.0 and 32.0 kg/m2 (inclusive)
* Women of childbearing potential (WOCBP) must have a negative pregnancy test and must not be lactating.
* Participants must agree to use an approved method(s) of highly effective contraception as defined in the protocol.

Exclusion Criteria:

* Clinically significant history or presence of gastrointestinal, hepatic, renal, cardiovascular, respiratory, endocrine, neurologic, hematologic, metabolic, autoimmune, or oncologic disorders that may affect safety or study outcomes.
* Chronic or active respiratory disease (e.g., asthma, COPD) or history of angioedema within 3 years.
* Active or chronic liver disease, or abnormal liver function tests (ALT, AST, or bilirubin outside reference range, except Gilbert's syndrome).
* QTcF >450 msec (males) or >470 msec (females).
* Renal impairment (creatinine clearance <90 mL/min) or thrombocytopenia (<150 × 10⁹/L).
* Positive test for hepatitis B surface or core antigen, hepatitis C (unless HCV-RNA negative), or HIV.
* Active respiratory infection within 5 days before study start.
* Recent or concurrent use of medications, herbal supplements, vaccines, or blood products that could interfere with study safety or interpretation.
* Participation in another investigational study within 30 days, or blood donation >400 mL within 30 days.
* Parts A and B only: Regular smoking (≥1 day per week) within 6 months prior to dosing, or a positive urine cotinine test at screening or Day -1.
* Excessive alcohol consumption (>21 drinks/week for males or >14 for females).
* History of severe drug reaction or anaphylaxis.
* Contraindication to, or unwillingness to undergo, bronchoscopy.
* Any psychiatric or medical condition that, in the investigator's opinion, could compromise safety or compliance.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-01-22 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Number and frequency of treatment-emergent adverse events (TEAEs) | From Day 1 until the end of the study (Day 85 for Part A; Day 106 for Parts A and B)
  To assess the safety and tolerability of single and multiple doses of RB042 when administered via a nebuliser to healthy adult volunteers and healthy adult smokers

SECONDARY OUTCOMES:
Maximum concentration (Cmax) | From Day 1 until the end of the study (Day 85 for Part A; Day 106 for Parts A and B)
  To characterize the Cmax of RB042 following single and multiple doses of RB042 administered via a nebuliser to healthy adult volunteers and healthy adult smokers
Time to maximum concentration (Tmax) | From Day 1 until the end of the study (Day 85 for Part A; Day 106 for Parts A and B)
  To characterize the Tmax of RB042 following single and multiple doses of RB042 administered via a nebuliser to healthy adult volunteers and healthy adult smokers
Terminal elimination half-life (t½) | From Day 1 until the end of the study (Day 85 for Part A; Day 106 for Parts A and B)
  To characterize the t½ of RB042 following single and multiple doses of RB042 administered via a nebuliser to healthy adult volunteers and healthy adult smokers
Area under the concentration-time curve (AUC) | From Day 1 until the end of the study (Day 85 for Part A; Day 106 for Parts A and B)
  To characterize the AUC of RB042 following single and multiple doses of RB042 administered via a nebuliser to healthy adult volunteers and healthy adult smokers
Trough concentration | On Days 7, 14, and 21
  To characterize the AUC of RB042 following multiple doses of RB042 administered via a nebuliser to healthy adult volunteers and healthy adult smokers

CONTACTS AND LOCATIONS:
Locations (1):
- Linear Clinical Research, Nedlands, Western Australia, Australia

IPD SHARING:
Plan to Share IPD: No